CLINICAL TRIAL: NCT00793585
Title: A Prospective, Randomized Controlled Study of Uric Acid on the Progression of IgA Nephropathy
Brief Title: A Controlled Study of Uric Acid on the Progression of IgA Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-PRGIgAN-002
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2011-07-01 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: IgA Nephropathy
Keywords: IgA nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol (Experimental): Allopurinol group:allopurinol, 100-300mg/d according to the levels of Scr(serum creatinine) and UA(uric acid), for those Scr < 1.5mg/dl (133 umol/L) at the baseline, allopurinol was given 100 mg three times daily.Patients diagnosed with hypertension received antihypertensive drugs with titration of CCB and β-blocker during the follow-up.The target of BP is less than 130/80mmHg.
  Interventions: Drug: allopurinol
- Control group (Other): Control group:(patient in this group were received health education and were encouraged to adhere to a low-purine diet and continue their usual therapy.Patients diagnosed with hypertension received antihypertensive drugs with titration of CCB and β-blocker during the follow-up.The target of BP is less than 130/80mmHg.
  Interventions: Other: continue their usual therapy

INTERVENTIONS:
Drug: allopurinol — Patients will receive the lifestyle modification and treatment of allopurinol (300 mg /d) and lifestyle modification for 4 weeks; when the UA level < 6mg/dl , the dosage changed to 200mg/d.
  Arms: Allopurinol
Other: continue their usual therapy — Patients will receive lifestyle modification and continue their usual therapy.
  Arms: Control group

SUMMARY:
This prospective, randomized controlled study will evaluate the effect of uric acid on the progression of IgA nephropathy.

DETAILED DESCRIPTION:
It has been reported that hyperuricemia is a risk factor for progression of IgAN. This will be a prospective, randomized study. Eligible IgAN patients will be randomized into the treatment group and the control group. Patients in treatment group will receive allopurinol and usual therapy. Patients in control group will receive usual therapy with placebo. If with hypertension, add the CCB and the β-blocker. Fasting uric acid, serum creatinine, albumin, routine blood test, urine microscopy and dipstick, proteinuria of 24 hours and blood pressure will be measured every month. After followed-up for 6 months, the curative effect of Allopurinol on blood pressure, proteinuria and the progression of IgA nephropathy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either sex, more than 18 years old, the range of age is 18 to 70 year old.
2. Biopsy-proven IgA nephropathy.
3. Proteinuria between 0.15g/d and 3.0g/d; and serum albumin level>3.5g/dl.
4. Serum creatinine < 3 mg/dl.
5. Uric acid > 6 mg//dl (360umol/dl) in female; Uric acid >7mg/dl (420umol/dl ) in male.
6. No history of taking ACEI or ARB within 2 weeks.
7. Blood pressure < 180/110 mmHg.
8. Subjects who agree to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Patients who have received prednisone or immunosuppressive drugs within 2 months.
2. Patients who must take ACEI or ARB due to other diseases.
3. Patients who have the history of allergy to allopurinol.
4. Unwillingness to follow the study protocol.
5. Active gout within 4 weeks.
6. Pregnancy or unwillingness to use contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, M.D. & Ph.D., Principal Investigator — 1st Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty hyperuricemic patients with IgA nephropathy were enrolled in the 1st affiliated hospital of sun yat-sen university between July 2007 and June 2008.
Pre-assignment Details: 323 primary IgAN patients were screened for enrollment according to inclusion criteria.
Groups:
- Control Group: Control group:(patient in this group were received health education and were encouraged to adhere to a low-purine diet.Patients diagnosed with hypertension received antihypertensive drugs with titration of CCB and β-blocker during the follow-up.The target of BP is less than 130/80mmHg.
- Allopurinol Group: Patients in the treatment group received allopurinol, 100-300mg/d according to the levels of Scr and UA. For those with Scr<1.5mg/dl (133µmol/L) at the baseline, allopurinol was given 100mg three times daily, and changed to 100mg twice daily when serum uric acid deceased to the normal range. For patients with Scr>=1.5mg/dl at baseline, allopurinol was initiated at 100mg twice daily and was decreased to 100mg daily when uric acid decreased into the normal range.
Period: Overall Study
Arm/Group | Control Group | Allopurinol Group
Started | 19 | 21
Completed | 17 | 18
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Allopurinol Group | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 21 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (10.3) | 39.7 (10.0) | 39.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 9 | 13 | 22
Region of Enrollment [Number; unit: participants]
  China | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Renal Function as Measured With eGFR
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: eGFR(min/ml)
Arm/Group | Control Group | Allopurinol Group
Number analyzed (Participants) | 19 | 21
eGFR(min/ml) | 68.9 (36.6) | 73.2 (34.8)

2. Secondary Outcome: The Longitudinal Change in Proteinuria and Blood Pressure(Including Changes in Antihypertensive Drugs Dosing).
Time Frame: baseline and 6 months
Population: We analysed all patient's data according to the ITT rule.And used the LOCF as the imputation technique.
Measure: Mean (Standard Deviation); unit: Upro/cr (mg/g)
Arm/Group | Control Group | Allopurinol Group
Number analyzed (Participants) | 19 | 21
Upro/cr (mg/g) | 1170.4 (951.9) | 1219.3 (1063.6)

ADVERSE EVENTS:
Arm/Group | Control Group | Allopurinol Group
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes